CLINICAL TRIAL: NCT06632002
Title: A Randomized, Double-blind, Non-inferiority Trial of a New Diabetes-specific Formula Compared to an Existing Diabetes-specific Formula on Nutritional Outcomes in Individuals With Diabetes Who Require Nutritional Support
Brief Title: Diabetes-specific Formulas on Nutritional Outcomes in Individuals With Diabetes Who Require Nutritional Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BL80
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Product (Experimental)
  Interventions: Other: DSF1; Other: Standard of Care (SOC)
- Control Product (Other)
  Interventions: Other: DSF2; Other: Standard of Care (SOC)

INTERVENTIONS:
Other: DSF1 — 220 mL
  Arms: Experimental Product
Other: DSF2 — 220 mL
  Arms: Control Product
Other: Standard of Care (SOC) — Standard of care

SUMMARY:
The study aims to demonstrate the non-inferiority of diabetes-specific formula (DSF)1 compared to DSF2 in individuals with type 1 diabetes, type 2 diabetes or prediabetes and who are at nutritional risk.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel, non-inferiority study. Eligible participants will be randomly allocated (at 1:1 ratio) to one of two groups: DSF1 (experimental group) or DSF2 (control group). Both groups will incorporate one serving of the DSF into their daily diet, in addition to receiving standard of care for diabetes. The total expected duration of the study is up to 104 days, including a run-in period of up to 14 days, followed by an intervention period of 90 days. At Day 1, participants will be randomized into one of the two groups (n = 50 per group): DSF1 or DSF2. Participants will start the intervention on Day 1 and complete the intervention on Day 90.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Has any of the following types of diabetes:

   1. Type 1 diabetes
   2. Type 2 diabetes
   3. Prediabetes
2. Has MNA-SF score of ≤ 11
3. Serum albumin less than 4.0 g/dL
4. Energy or protein intake less than recommended
5. BMI less than 30.0 kg/m2
6. Either a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to the study
7. Female of childbearing potential to use an effective method of birth control
8. Chronic medication type and dose to be constant and maintained throughout the study
9. Willing to follow the protocol throughout the study
10. At least a two-week washout period between the completion of a previous research study and start in current study
11. Willing to refrain from taking non-study diabetes-specific formula over the course of the study.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Has a screening HbA1c level less than 5.0% or ≥ 10%
2. Has a current infection, inpatient surgery or received systemic corticosteroid treatment in the last 3 months; or received antibiotics in the last 3 weeks
3. Has active malignancy within the last 5 years
4. Has significant cardiovascular event within 6 months prior to the study or history of congestive heart failure
5. Has end-stage organ failure or is post-organ transplant
6. Has current or history of renal disease or on dialysis or severe gastroparesis
7. Has current hepatic disease
8. Has a recent acute infection, physiologic stress or trauma within 1 month prior to the study
9. Has had bariatric surgery including gastric balloon; history of gastrointestinal disease or intestinal surgery that can interfere with consumption or digestion or absorption of study product
10. Has a chronic, contagious, infectious disease
11. Has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study procedures
12. Taking any herbals, dietary supplements or medications during the past 4 weeks prior to the study
13. Using diabetes-specific formula(s) or oral nutritional supplement formula(s) in more than one eating occasion per week within the past 3 months
14. Has clotting or bleeding disorders
15. Has blood or blood-related diseases
16. Has received blood transfusion within the last 3 weeks
17. Has allergy or intolerance to the study product
18. Anticipated poor compliance to the study as assessed by the Investigator
19. Participates in another study that has not been approved as a concomitant study by Abbott Nutrition

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Serum albumin | Study Day 1 to Day 90
  Change in serum albumin levels from baseline to Day 90

SECONDARY OUTCOMES:
Serum albumin | Study Days 45 and 90
  Serum albumin levels
Malnutrition risk | Study Days 45 and 90
  Mini Nutritional Assessment - Short Form (MNA®-SF) a validated screening tool for identifying elderly persons who are at risk for malnutrition, or who are already malnourished. It classifies participants into one of three categories:
  1. Normal nutritional status/score =12 to 14 points,
  2. At risk of malnutrition/score = 8 to 11 points,
  3. Malnourished/score = 0 to 7 points. Minimum point = 0, Maximum points = 14. Lower score indicates worse outcome, i.e., at risk of malnutrition or malnourished.
Malnutrition risk | Study Days 45 and 90
  Malnutrition Universal Screening Tool (MUST) is a widely used screening tool for malnutrition. It classifies participants into one of three nutrition status categories:
  1. Low risk/score = 0,
  2. Medium risk/score = 1,
  3. High risk/score ≥ 2. Minimum value = 0, Maximum value = 6. Higher score indicates worse outcome, i.e., increased risk of malnutrition.
Serum prealbumin | Study Days 45 and 90
  Serum prealbumin levels
Body weight | Study Days 45 and 90
  Body weight measured in kg
Body mass index (BMI) | Study Days 45 and 90
  Calculated as weight (kg)/height (m)2
Mid arm circumference | Study Days 45 and 90
  Mid arm circumference measured in cm
Mid arm muscle circumference | Study Days 45 and 90
  Mid arm muscle circumference measured in cm
Triceps skinfold thickness | Study Days 45 and 90
  Triceps skinfold thickness measured in mm
Calf circumference | Study Days 45 and 90
  Calf circumference measured in cm
Waist circumference | Study Days 45 and 90
  Waist circumference measured in cm
Hip circumference | Study Days 45 and 90
  Hip circumference measured in cm
Waist-to-hip-ratio | Study Days 45 and 90
  Waist-to-hip-ratio
Hemoglobin A1c (HbA1c) | Study Days 45 and 90
  HbA1c levels
Fasting plasma glucose | Study Days 45 and 90
  Fasting plasma glucose levels
2-hour postprandial glucose | Study Days 45 and 90
  2-hour postprandial glucose levels
Glycated albumin | Study Days 45 and 90
  Glycated albumin levels
Triglycerides | Study Days 45 and 90
  Triglycerides levels
High density lipoprotein (HDL) cholesterol | Study Days 45 and 90
  HDL cholesterol levels
Low density lipoprotein (LDL) cholesterol | Study Days 45 and 90
  LDL cholesterol levels

OTHER OUTCOMES:
Energy, macronutrient and micronutrient intakes | Study Days 45 and 90
  A 3-day Dietary Record (two weekdays and one weekend day) will be completed by participant for the week prior Study Day 45 and 90 and evaluated by a dietitian. Nutrient analysis will be performed using a dietary analysis program.
Energy, macronutrient and micronutrient adequacy | Study Days 45 and 90
  Nutrient adequacy will be determined by comparing nutrient intakes (outcome No. 21) against sex- and age- specific local recommended nutrient intakes (RNI).
Product intake compliance | Study Days 90
  Compliance to study product prescribed over 90-day intervention period
Adverse events | Study Day 1 to Day 90
  Reported adverse events for assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Yen Ling Ow, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No